CLINICAL TRIAL: NCT01490918
Title: A Multicenter, Randomized, Double Blind, Placebo-controlled Study to Evaluate the Efficacy of Acarbose Added on Top of Metformin and Sitagliptin Combination Treatment in Type 2 Diabetes Mellitus Patients
Brief Title: Study to Evaluate the Efficacy of Acarbose,Metformin,Sitagliptin Combination Treatment in DM Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Kun-Ho Yoon, Professor, Medical doctor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACADEMIC
Record Dates: First submitted 2011-12-09; First posted 2011-12-13 (Estimated); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Acarbose; ACADEMIC
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acarbose; Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: placebo medication
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acarbose placebo, Metformin, Sitagliptin (Placebo Comparator): The Acarbose placebo should be changed into real Acarbose from the 16th week.
  Interventions: Drug: Placebo acarbose
- Sitagliptin, Metformin, Acarbose (Experimental): Metformin, Sitagliptin, Acarbose group
  Interventions: Drug: Acarbose
- Metformin placebo, Sitagliptin, Acarbose (Other): The Metformin placebo should be changed into real Metformin from the 16th week.
  Interventions: Drug: placebo metformin

INTERVENTIONS:
Drug: Acarbose — Acarbose 50mg b.i.d at first, at the 2nd week 50mg t.i.d and the 4th week, 100mg tid.
  Other Names: triple combination
  Arms: Sitagliptin, Metformin, Acarbose
Drug: Placebo acarbose — acarbose placebo
  Other Names: dual combination (metformin+sitagliptin)
  Arms: Acarbose placebo, Metformin, Sitagliptin
Drug: placebo metformin — metformin placebo
  Other Names: dual combination (acarbose + sitagliptin)
  Arms: Metformin placebo, Sitagliptin, Acarbose

SUMMARY:
Primary objective To evaluate the efficacy of Acarbose add-on therapy on glucose control in subjects with type 2 diabetes inadequately controlled with Metformin and Sitagliptin combination therapy.

The effect of acarbose, an alpha glucosidase inhibitor as a third-line therapeutic medication in subject who are inadequately controlled with metformin and DPP4 inhibitor will be evaluated with multicenter, randomized, 24-week, double blinded, placebo-controlled study in Korea.

DETAILED DESCRIPTION:
Eligible subjects will be assigned among 3 groups randomly at a ration of 2:2:1 to the following groups and primary efficacy variable analyzed at week 16.

group 1 : acarbose placebo + metformin + sitagliptin (with switching placebo to acarbose qt week 16) group 2 : acarbose + metformin + sitagliptin group 3 : acarbose + metformin placebo + sitagliptin (with switching placebo to metformin at week 16)

After 16 week of treatment, all subjects in 3 groups will be treated as triple combination of acarbose + metformin + sitagliptin, and diabetes related variables be collected and analyzed.

1. Primary Endpoint Changes in HbA1c (hemoglobin A1c) at 16 week from baseline between group1 vs grou2
2. Secondary Endpoints (1) Changes of HbA1c at 24 week between 3 groups (2) Changed of post-prandial blood glucose at 2 hour (ppg2h) at 16, 24 week

for exploratory purpose, following data will be collected and analyzed

1. continuous glucose monitoring system (CGMS) data among selected subjects in 3 groups
2. mixed meal tolerance test in only available institution. (glucose, insulin, GLP-1, GIP, glucagon ) among selected subjects in group 1 and group 2
3. oxidative stress markers (8-OHdG, nitrotyrosin, CML)
4. self monitoring of blood glucose

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with type-II diabetes mellitus;
2. Subjects aged between 20 and 80;
3. Subjects whose HbA1c ratio is between 7.0% and 10.0%;
4. Subjects who took Metformin and Sitagliptin for at least 12 weeks;
5. Subjects who were given the explanation about this clinical study and signed the consent form.

Exclusion Criteria:

1. Subjects who have taken drugs that are likely to affect blood glucose or who need to take such drugs, e.g., glucocorticoid;
2. Subjects with severe renal diseases (men: Scr>1.5 / women: Scr>1.4);
3. Subjects with severe liver diseases or whose AST and ALT are at least 2.5 times higher than the upper limits of normal (ULN);
4. Subjects having the case history of lactic acidosis;
5. Subjects who have the case history of myocardial infarction or unstable angina or who underwent the coronary artery bypass graft 6 months before the screening test or who have arrhythmia to be treated;
6. Subjects with congestive heart failures to be treated;
7. Subjects who fall into New York Heart Association (NYHA) class III or IV;
8. Subjects having the case history of acute or chronic metabolic acidosis including ketoacidosis;
9. Subjects who have been pregnant or who are in the period of lactation;
10. Subjects diagnosed with malignant tumors within 5 years;
11. Subjects who are hypersensitive to Metformin, Sitagliptin and Acarbose or their ingredients;
12. Subjects with inflammatory bowel diseases or intestinal ulcers or enterostenosis (includes Subjects who are vulnerable to enterostenosis) or chronic enteric diseases related to digestion and absorption or whose symptoms are likely to worsen due to intestinal gas;
13. Subjects who participated in other clinical studies as Subjects within 60 days before this study (or before taking the investigational drugs);
14. Subjects judged unfit for this study by investigators.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2012-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kun-HO Yoon, professor, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- MedicalExcellence, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Acarbose Placebo, Metformin, Sitagliptin: Metformin and sitagliptin and placebo treatment for 16 weeks. Placebo was changed to acarbose at 16 week and maintained for another 8 weeks.
- Sitagliptin, Metformin, Acarbose: Metformin and sitagliptin and acarbose treatment for 24 weeks.
- Metformin Placebo, Sitagliptin, Acarbose: Placebo and sitagliptin and acarbose treatment for 16 weeks. Placebo was changed to acarbose at 16 week and maintained for another 8 weeks. The Metformin placebo should be changed into real Metformin from the 16th week.
Period: Overall Study
Arm/Group | Acarbose Placebo, Metformin, Sitagliptin | Sitagliptin, Metformin, Acarbose | Metformin Placebo, Sitagliptin, Acarbose
Started | 65 | 66 | 34
Completed | 52 | 52 | 22
Not Completed | 13 | 14 | 12
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 8 | 3
Not completed — Adverse Event | 0 | 0 | 1
Not completed — other cause | 4 | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Acarbose Placebo, Metformin, Sitagliptin: The dose of Acarbose should be 50mg b.i.d, 50mg t.i.d and 100mg t.i.d at the 18th week, the 20th week and the 24th week respectively. The Acarbose placebo should be changed into real Acarbose from the 16th week.
  Acarbose: The dose of Acarbose or its placebo should be 50mg b.i.d at first. At the 2nd week and the 4th week, it should be 50mg t.i.d and 100mg t.i.d respectively
- Sitagliptin, Metformin, Acarbose: The group's drugs not include placebo. (Metformin, Sitagliptin, Acarbose)
  Acarbose: The dose of Acarbose or its placebo should be 50mg b.i.d at first. At the 2nd week and the 4th week, it should be 50mg t.i.d and 100mg t.i.d respectively
- Metformin Placebo, Sitagliptin, Acarbose: The Metformin placebo should be changed into real Metformin from the 16th week.
  Acarbose: The dose of Acarbose or its placebo should be 50mg b.i.d at first. At the 2nd week and the 4th week, it should be 50mg t.i.d and 100mg t.i.d respectively
- Total: Total of all reporting groups
Arm/Group | Acarbose Placebo, Metformin, Sitagliptin | Sitagliptin, Metformin, Acarbose | Metformin Placebo, Sitagliptin, Acarbose | Total
Number analyzed (Participants) | 65 | 66 | 34 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.55 (10.51) | 60.89 (8.8) | 60.15 (9.92) | 59.03 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 43 | 14 | 87
  Male | 35 | 23 | 20 | 78
Region of Enrollment [Number; unit: participants]
  South Korea | 65 | 66 | 34 | 165

OUTCOME MEASURES:

1. Primary Outcome: The Change of Glycated Hemoglogin(HbA1c) From Baseline to 16 Weeks of Treatment
Description: The change of glycated hemoglogin(HbA1c) from baseline to 16 weeks of treatment between Placebo + Metformin+Sitagliptin and Metformin + Sitagliptin + Acarbose group
Time Frame: baseline, 16 weeks
Population: ITT: intention to treatment, All subject randomized to each treatment group
Measure: Mean (Standard Error); unit: % of HbA1c
Groups:
- Placebo+Metformin+Sitagliptin: Metformin and sitagliptin and placebo treatment for 16 weeks. Placebo was changed to acarbose at 16 week and maintained for another 8 weeks as triple combination of acarbose + metformin + sitagliptin
- Sitagliptin+Metformin+Acarbose: Metformin and sitagliptin and acarbose treatment for 24 weeks.
- Placebo+Sitagliptin+Acarbose: Placebo and sitagliptin and acarbose treatment for 16 weeks. The placebo will be changed to Metformin from the 16th week and maintained another 8 week for triple combination of metformin + sitagliptin + acarbose.
Arm/Group | Placebo+Metformin+Sitagliptin | Sitagliptin+Metformin+Acarbose | Placebo+Sitagliptin+Acarbose
Number analyzed (Participants) | 65 | 66 | 34
% of HbA1c | -0.09 (0.1) | -0.44 (0.08) | 0.84 (0.21)
Statistical Analysis 1: Comparison: Placebo+Metformin+Sitagliptin vs Sitagliptin+Metformin+Acarbose; primary outcome efficacy will be evaluated between group 1(placebo + metfromin + sitagliptin) and 2 (sitagliptine + metformin + acarbose); Test type: Superiority; p = 0.0036, ANCOVA — The threshold for statistical significance was p=0.05; Baselin HbA1c as covariate

2. Secondary Outcome: The Change of HbA1c From Baseline to 24 Weeks of Treatment
Description: The change of glycated hemoglogin(HbA1c) from baseline to 24 weeks of treatment between 3 groups
Time Frame: baseline, 24 weeks
Population: ITT: intention to treatment, All subject randomized to each treatment group
Measure: Mean (Standard Deviation); unit: % of HbA1c
Arm/Group | Placebo+Metformin+Sitagliptin | Sitagliptin+Metformin+Acarbose | Placebo+Sitagliptin+Acarbose
Number analyzed (Participants) | 65 | 66 | 34
% of HbA1c | -0.34 (0.82) | -0.47 (0.78) | 0.23 (1.32)
Statistical Analysis 1: Comparison: Placebo+Metformin+Sitagliptin vs Sitagliptin+Metformin+Acarbose vs Placebo+Sitagliptin+Acarbose; Test type: Superiority; p < 0.0001, ANCOVA — The threshold for statistical significance was p=0.05; Baseline HbA1c as covariate

3. Secondary Outcome: The Change of PPG2hr From Baseline to 24 Weeks of Treatment
Description: The change of PPG2hr (post prandia blood glucose 2hr from baseline to 24 weeks of treatment between 3 groups
Time Frame: baseline, 24 weeks
Population: ITT: intention to treatment, All subject randomized to each treatment group
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Placebo+Metformin+Sitagliptin: Metformin and sitagliptin and placebo treatment for 16 weeks. Placebo was changed to acarbose at 16 week and maintained for another 8 weeks.
- Placebo+Sitagliptin+Acarbose: Placebo and sitagliptin and acarbose treatment for 16 weeks. Placebo was changed to acarbose at 16 week and maintained for another 8 weeks. The Metformin placebo should be changed into real Metformin from the 16th week.
Arm/Group | Placebo+Metformin+Sitagliptin | Sitagliptin+Metformin+Acarbose | Placebo+Sitagliptin+Acarbose
Number analyzed (Participants) | 63 | 66 | 34
mmol/L | -1.73 (3.38) | -1.76 (3.53) | 0.06 (4.53)
Statistical Analysis 1: Comparison: Placebo+Metformin+Sitagliptin vs Sitagliptin+Metformin+Acarbose vs Placebo+Sitagliptin+Acarbose; Test type: Superiority; p = 0.0185, ANCOVA — The threshold for statistical significance was p=0.05; baseline PPG2hr as covariate

4. Secondary Outcome: Changes in Glucose During Meal Tolerance Test Between 2 Group(Group 1 vs Group 2),
Description: Change of AUC(area under the curve) of glucose at 16 week from baseline between 2 groups (placebo+metformin + sitagliptin vs acarbose + metformin + sitagliptin)
Time Frame: Visit 2(baseline) and Visit 5(16W)
Measure: Mean (Standard Deviation); unit: mg min/dL
Arm/Group | Placebo+Metformin+Sitagliptin | Sitagliptin+Metformin+Acarbose
Number analyzed (Participants) | 12 | 13
mg min/dL | 28.85 (2168.64) | -743.08 (1278.28)
Statistical Analysis 1: Comparison: Placebo+Metformin+Sitagliptin vs Sitagliptin+Metformin+Acarbose; Test type: Superiority; p = 0.0356, ANCOVA — The threshold for statistical significance was p=0.05; baseline data as covariate

5. Secondary Outcome: Changes in Insulin During Mixed Meal Tolerance Test Between 2 Group(Group 1 vs Group 2),
Description: Change of AUC(area under the curve) of insulin at 16 week from baseline between 2 groups (placebo+metformin + sitagliptin vs acarbose + metformin + sitagliptin)
Time Frame: Visit 2(baseline) and Visit 5(16W)
Measure: Mean (Standard Deviation); unit: pg min/mL
Arm/Group | Placebo+Metformin+Sitagliptin | Sitagliptin+Metformin+Acarbose
Number analyzed (Participants) | 13 | 12
pg min/mL | 647.65 (3854.75) | 221.42 (8339.6)
Statistical Analysis 1: Comparison: Placebo+Metformin+Sitagliptin vs Sitagliptin+Metformin+Acarbose; Test type: Superiority; p = 0.8258, ANCOVA — The threshold for statistical significance was p=0.05; baseline data as covariate

6. Secondary Outcome: Change in Active GLP-1 at 0 Minute During Mixed Meal Test Between 2 Groups (Group 1, group2)
Description: Change of active GLP-1 at 0 minute during mixed meal test at 16 week from baseline between 2 groups(group1, group2)
Time Frame: baseline, 16 week
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Placebo+Metformin+Sitagliptin | Sitagliptin+Metformin+Acarbose
Number analyzed (Participants) | 12 | 13
pg/ml | -8.55 (19.01) | -9.33 (31.12)
Statistical Analysis 1: Comparison: Placebo+Metformin+Sitagliptin vs Sitagliptin+Metformin+Acarbose; Test type: Superiority; p = 0.9217, ANCOVA — The threshold for statistical significance was p=0.05; baseline data as covariate

7. Secondary Outcome: Change in Active GLP-1 at 120 Minute During Mixed Meal Test Between 2 Groups (Group 1, group2)
Description: Change of active GLP-1 at 120 minute during mixed meal test at 16 week from baseline between 2 groups(group1, group2)
Time Frame: baseline, 16 week
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Placebo+Metformin+Sitagliptin | Sitagliptin+Metformin+Acarbose
Number analyzed (Participants) | 12 | 13
pg/ml | -32.92 (21.78) | -23.36 (33.43)
Statistical Analysis 1: Comparison: Placebo+Metformin+Sitagliptin vs Sitagliptin+Metformin+Acarbose; Test type: Superiority; p = 0.16, ANCOVA — The threshold for statistical significance was p=0.05; baseline data as covariate

8. Secondary Outcome: Changes in Glucagon During Meal Tolerance Test Between 2 Group(Group 1 vs Group 2),
Description: Change of AUC(area under the curve) of glucagon at 16 week from baseline between 2 groups (placebo+metformin + sitagliptin vs acarbose + metformin + sitagliptin)
Time Frame: Visit 2(baseline) and Visit 5(16W)
Measure: Mean (Standard Deviation); unit: min pg/mL
Arm/Group | Placebo+Metformin+Sitagliptin | Sitagliptin+Metformin+Acarbose
Number analyzed (Participants) | 9 | 9
min pg/mL | -79.22 (833.59) | -1411.79 (1049.41)
Statistical Analysis 1: Comparison: Placebo+Metformin+Sitagliptin vs Sitagliptin+Metformin+Acarbose; Test type: Superiority; p = 0.004, ANCOVA — The threshold for statistical significance was p=0.05; baseline data as covariate

9. Other Pre Specified Outcome: Changes in Mean Glucose During CGMS Between 3 Group
Description: Change of mean glucose of CGMS(continuous glucose monitoring system) data at 16 week from baseline between 3 groups
Time Frame: Visit 2(baseline) and Visit 5(16W)
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Placebo + Sitagliptin + Acarbose: Placebo and sitagliptin and acarbose treatment for 16 weeks. The placebo will be changed to Metformin from the 16th week and maintained another 8 week for triple combination of metformin + sitagliptin + acarbose.
Arm/Group | Placebo+Metformin+Sitagliptin | Sitagliptin+Metformin+Acarbose | Placebo + Sitagliptin + Acarbose
Number analyzed (Participants) | 11 | 13 | 6
mmol/L | -0.91 (0.81) | -1.16 (0.49) | 3.22 (1.25)
Statistical Analysis 1: Comparison: Placebo+Metformin+Sitagliptin vs Sitagliptin+Metformin+Acarbose vs Placebo + Sitagliptin + Acarbose; Test type: Superiority; p = 0.292, ANCOVA — The threshold for statistical significance was p=0.05; baseline data as covariate

10. Other Pre Specified Outcome: Changes in Variation of Glucose During CGMS Between 3 Group
Description: Change of standard deviation of CGMS(continuous glucose monitoring system) data at 16 week from baseline between 3 groups (placebo+metformin + sitagliptin vs acarbose + metformin + sitagliptin vs placebo + acarbose + sitagliptin)
Time Frame: Visit 2(baseline) and Visit 5(16W)
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Placebo + Acarbose + Sitagliptin: Placebo and sitagliptin and acarbose treatment for 16 weeks. The placebo will be changed to Metformin from the 16th week and maintained another 8 week for triple combination of metformin + sitagliptin + acarbose.
Arm/Group | Placebo+Metformin+Sitagliptin | Sitagliptin+Metformin+Acarbose | Placebo + Acarbose + Sitagliptin
Number analyzed (Participants) | 11 | 13 | 6
mmol/L | -0.33 (1.0) | -0.65 (0.8) | 0.03 (0.29)
Statistical Analysis 1: Comparison: Placebo+Metformin+Sitagliptin vs Sitagliptin+Metformin+Acarbose vs Placebo + Acarbose + Sitagliptin; Test type: Superiority; p = 0.314, ANCOVA — The threshold for statistical significance was p=0.05; baseline data as covariate

11. Other Pre Specified Outcome: Changes in MAGE of Glucose During CGMS Between 2 Group(Group 1 vs Group 2),
Description: Change of mean amplitude of glycemic excursion of CGMS(continuous glucose monitoring system) data at 16 week from baseline between 2 groups (placebo+metformin + sitagliptin vs acarbose + metformin + sitagliptin)
Time Frame: Visit 2(baseline) and Visit 5(16W)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo+Metformin+Sitagliptin | Sitagliptin+Metformin+Acarbose | Placebo + Acarbose + Sitagliptin
Number analyzed (Participants) | 11 | 13 | 6
mg/dL | -8.79 (15.01) | -18.5 (13.23) | 2.72 (2.72)
Statistical Analysis 1: Comparison: Placebo+Metformin+Sitagliptin vs Sitagliptin+Metformin+Acarbose vs Placebo + Acarbose + Sitagliptin; Test type: Superiority; p = 0.7563, ANCOVA — The threshold for statistical significance was p=0.05; baseline data as covariate

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: total number afffected by any other adverse event : included SAEs
Arm/Group | Acarbose Placebo, Metformin, Sitagliptin | Sitagliptin, Metformin, Acarbose | Metformin Placebo, Sitagliptin, Acarbose
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/66 | 0/34
Serious Adverse Events (participants affected / at risk) | 2/65 | 1/66 | 0/34
Other Adverse Events (participants affected / at risk) | 14/65 | 19/66 | 11/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acarbose Placebo, Metformin, Sitagliptin (N=65) | Sitagliptin, Metformin, Acarbose (N=66) | Metformin Placebo, Sitagliptin, Acarbose (N=34)
chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acarbose Placebo, Metformin, Sitagliptin (N=65) | Sitagliptin, Metformin, Acarbose (N=66) | Metformin Placebo, Sitagliptin, Acarbose (N=34)
cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
dyspepsia (Gastrointestinal disorders) | 2 (2) | 6 (6) | 0 (0)
flatulence (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
large intestinal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
toothcache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
nasopharyngitis (Infections and infestations) | 1 (1) | 2 (3) | 1 (1)
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ALT increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
AST increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
diabetes mellitus inadequate controll (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4)
hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2)
lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
uterine leimyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
prorteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Evaluation of GIP and oxidative stress markers (8-OHdG, Nitrotyrosin) were not analyzed due to limited number of sample and technical problems leading to uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No